CLINICAL TRIAL: NCT06212960
Title: Double-blind, Randomized, Parallel Design, Active-controlled Phase 1 Clinical Trial to Evaluate the Efficacy and Safety of DWP712 and Botox® in Adult Patients in Need of Moderate to Severe Glabellar Lines
Brief Title: Evaluate the Safety and Explore the Efficacy of DWP712 With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP712101
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-01

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP712 (Experimental): Patients were intramuscularly injected (IM) with a total of 20U of DWP712 in 5 places of 0.1 mL (4 U/0.1 mL) each on the glabellar line.
  Interventions: Biological: DWP712
- Botox® (Active Comparator): Patients were intramuscularly injected (IM) with a total of 20U of BOTOX® in 5 places of 0.1 mL (4 U/0.1 mL) each on the glabellar line.
  Interventions: Biological: BOTOX®

INTERVENTIONS:
Biological: DWP712 — Clostridium botulinum Toxin
  Arms: DWP712
Biological: BOTOX® — Clostridium botulinum Toxin
  Arms: Botox®

SUMMARY:
To evaluate the safety of 12-week administration of DWP712 inj. in subjects with moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with facial wrinkle scale (FWS) score of visual appearance of glabellar lines ≥2 (moderate) at maximum frown as assessed by the investigator at screening

Exclusion Criteria:

-

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Number of occurrences for grade 3 or higher adverse drug reactions (ADRs) according to CTCAE 5.0 | At 4, 8, 12 week after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, MD, Ph.D, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No